CLINICAL TRIAL: NCT00725439
Title: An Open Label Pilot Trial to Assess the Safety and Efficacy of Oral R115866 in the Treatment of Moderate to Severe Facial Acne
Brief Title: An Open Label Trial to Assess the Safety and Efficacy of Oral R115866 in the Treatment Facial Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT0700BEL001
Record Dates: First submitted 2008-07-17; First posted 2008-07-30 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — R 115866

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Talarozole
  Interventions: Drug: Talarozole

INTERVENTIONS:
Drug: Talarozole — Oral Dose 1.0 mg once daily
  Other Names: Rambazole; R115866

SUMMARY:
This study is looking at a new oral drug to treat acne. All patients in the study will get active drug, there is no placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Presence of moderate to severe facial acne vulgaris: having a minimum of 15 papules and/or pustules and at least 2 nodulocystic lesions
* In good general health and free of any disease state or physical condition which, in the investigator's opinion, might have impaired evaluation of acne or exposed the subject to an unacceptable risk by trial participation

Exclusion Criteria:

* Subjects with types of acne other than acne vulgaris
* Significant coexisting hepatic, renal, or bone marrow disease, hyperlipidemia, chronic pancreatitis, osteoporosis, or a history indicating adrenal cortex dysfunction or any other serious disease (including cancer and subjects known to be HIV positive)
* History of any malignancy in the past 5 years, except for adequately treated basal cell carcinoma of the skin
* History of heart failure, myocardial infarction within the past six months, cardiac arrhythmia, or under treatment for heart disorders
* Clinically significant abnormal ECG-intervals or morphology of the ECG; QT or QTc >470 ms in females or >450 ms in males
* Use of vitamin A (>1000 microgram/day), phenytoin, carbamazepine, warfarin, rifampicin, tetracyclines, ketoconazole, itraconazole, astemizole, terfenadine, cisapride, anti-psychotics, anti-depressants, lithium, antimalarials, alpha-blocking drugs, angiotensin-converting enzyme inhibitors, cyclosporin A, glucocorticosteroids and non-steroid anti-inflammatory drugs, non-potassium-sparing diuretics
* Use of oral retinoids 6 months prior to Visit 1
* Use of other oral/topical therapy for acne unless stopped at Visit 1
* Use of ultraviolet light (including artificial UVA and UVB as well as excessive natural sun exposure) unless stopped at Visit 1

Ages: 16 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Facial Lesion Count | Post 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. D. Roseeuw, MD, Principal Investigator — Department Dermatology, University Hospital Brussel (UZ Brussel)
Locations (3):
- Belgium (2):
  - Department of Dermatology, UZ Brussel, Brussels
  - Private Practice in Dermatology, Vilvoorde
- Albert Schweitzer Hospital, Dermatology, Zwijndrecht, Netherlands